CLINICAL TRIAL: NCT05913674
Title: Technical Feasibility of Modified Early Post-Operative Intraperitoneal Chemotherapy (mEPIC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CER-CEMTL 2023-3236
Record Dates: First submitted 2023-05-25; First posted 2023-06-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Peritoneal Carcinomatosis; Appendiceal Neoplasms; Colorectal Cancer Metastatic
Keywords: Intraperitoneal chemotherapy; Early post-operative intraperitoneal chemotherapy; Fluorouracil; Hyperthermic intraperitoneal chemotherapy; Cytoreductive surgery; mEPIC
MeSH Terms: conditions — Peritoneal Neoplasms; Appendiceal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mEPIC (Experimental): Adults (male and female) with a diagnosis of appendicular or colorectal cancer with peritoneal carcinomatosis will undergo mEPIC on post-operative days 1 and 2 following cytoreductive surgery and hyperthermic intraperitoneal chemotherapy.
  Interventions: Drug: Modified early post-operative intraperitoneal chemotherapy (mEPIC)

INTERVENTIONS:
Drug: Modified early post-operative intraperitoneal chemotherapy (mEPIC) — On post-operative days 1 and 2, an abdominal reservoir is obtained by administering 1000 mL of plasmalyte with 50 mEq NaHCO3 via a Tenckhoff catheter. Participants will then receive an intraperitoneal fluorouracil bolus of 400 mg/m2 administered over 1 to 2 minutes followed by a continuous intraperitoneal fluorouracil infusion of 1200 mg/m2 over the next 24 hours. During the continuous intraperitoneal infusion of fluorouracil, 50 mg of folinic acid is administered intravenously.
  After completion of mEPIC day 1, the perfusate is drained out before starting mEPIC day 2.
  Other Names: mEPIC

SUMMARY:
The goal of this prospective phase II unicentric Canadian clinical trial is to clarify the feasibility of modified early post-operative intraperitoneal chemotherapy (mEPIC) following cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) in the clinical context of peritoneal carcinomatosis from colorectal and appendicular neoplasms.

The primary objective of this study is to confirm the feasibility of mEPIC by evaluating its completion rate compared to the one of historical standard early post-operative intraperitoneal chemotherapy (EPIC) cohorts. The secondary objectives of the study are to evaluate the safety of the mEPIC protocol by monitoring adverse events arising during the protocol and to assess logistical implementation barriers for the nursing and Oncology pharmacy teams, respectively.

Participants will undergo a modified schedule of EPIC (mEPIC) designed to maximize therapeutic benefit by exploiting the known pharmacokinetics and pharmacodynamics properties of fluorouracil (5-FU) while limiting the logistical issues of the standard protocol. mEPIC consists in shortening the original protocol from five to two days of postoperative intraperitoneal chemotherapy. Additionally, instead of solely administering a singular 5-FU bolus per 24 hours-period, mEPIC is based on the De Gramont intravenous regimen and consists of administering one intraperitoneal bolus of 5-FU (400 mg/m2) followed by a 24 hours-intraperitoneal infusion of 5-FU (1200 mg/m2) on postoperative days 1 and 2.

DETAILED DESCRIPTION:
Early postoperative intraperitoneal chemotherapy (EPIC) was first introduced by Sugarbaker in the 1990s in an effort to reduce disease recurrence and to prolong long-term survival of patients with peritoneal carcinomatosis from colorectal and appendicular malignancies including pseudomyxoma peritonei (PMP). Given the high risk of peritoneal recurrence, even after optimal cytoreduction, EPIC was a simple way of delivering high doses of cytotoxic agents targeted at the peritoneal surfaces without systemic compromise and eliminating any residual microscopic tumor deposits before the formation of fibrinous adhesions. The original protocol consists of administering 650 mg / m2 of intraperitoneal Fluorouracil (5-FU) in hypertonic, high molecular weight solution on postoperative days one to five. This solution is administered as an intraperitoneal bolus, remains for 23 hours with the surgical drains clamped before one hour of free drainage. Currently, there is no definitive randomised data comparing the benefit of EPIC versus no EPIC in any indication. One study that evaluated repeated cycles of intraperitoneal 5-FU in colon cancer demonstrated improved survival, but the study was discontinued early due to poor recruitment. Non-randomised data from the St George Hospital Peritoneal Surface Malignancy Program suggests a benefit for the addition of EPIC to hyperthermic intraperitoneal chemotherapy (HIPEC) with respect to survival outcomes in low-grade appendiceal cancers with no differences in morbidity but requires increased time in high dependency care unit. A recent study also demonstrates that in low-grade appendiceal neoplasms with pseudomyxoma peritonei, the addition of EPIC to HIPEC with cytoreductive surgery (CRS) improves overall survival in propensity score matched cases but results in prolonged hospitalisation. There is also conflicting data showing no advantage for the addition of EPIC to HIPEC in colorectal and high grade appendiceal cancer and an increased rate of grade III/IV complications.

From a therapeutic perspective, the use of intraperitoneal 5-FU benefits from the high peritoneal to plasma area under the curve, hence allowing the administration of higher intraperitoneal doses than intravenous doses with a resultant 250-fold increased tissue exposure. Even with significantly higher doses of 5-FU, systemic toxicities are much lower than systemic infusion due in part from the first pass metabolism through the liver. However, the standard EPIC protocol does not take into account the short perfusate half-life of 5-FU (0.75-1.5 hour). Consequently, by administering it as a large bolus, the majority of 5-FU is metabolized from the intraperitoneal compartment within 4-7.5 hours even though the solution remains intraperitoneally for 23 hours. In comparison to systemic therapy, infusions regimens of 5-FU based on protracted venous infusion or the so-called De Gramont regimen have essentially replaced bolus regimens such as the Mayo and Roswell Park regimens due to superior efficacy and better toxicity profiles. It consists in administering a bolus of 5-FU to achieve therapeutic concentrations followed by protracted venous infusion of 5-FU. This mode of administration also maximizes the inhibition of thymidylate synthase and other targets of 5-FU.

Additionally, there are clinical and administrative down-sides to the existing standard EPIC. These include: protracted occupancy of high dependency unit beds with a high nurse to patient ratio, which aggravates existing access issues. Furthermore, there are risks of abdominal tamponade, generalised discomfort during the procedure, prolonged ileus and increased risk of fistula and collection, hence prolonging length of stay. For these mentioned reasons, many patients do not complete every day of the planned treatment. For instance, out of the 435 patients who received EPIC in a high-volume center (St George Hospital) between 1996 and 2017, 269 (61.8%) completed the 5-day protocol, 33 (7.6%), 30 (6.9%), 45 (10.3%) and 58 (13.3%) completed 1, 2, 3 and 4 days of EPIC, respectively.

Rationale for Performing this Study:

Although, there is no randomised evidence to support EPIC, it has become one of the standard therapies for management of colorectal and appendicular neoplasms with peritoneal carcinomatosis in many high-volume surgical oncology centers. There is a need to devise a logistically more feasible regimen and also exploit the known pharmacokinetics and pharmacodynamics properties of 5-FU. Our phase II trial proposes a modified schedule of EPIC (mEPIC) designed to maximize therapeutic advantages and reduce logistical barriers. This modified EPIC (mEPIC) consists in shortening the original protocol from five to two days of postoperative intraperitoneal chemotherapy. Additionally, instead of solely administering a singular 5-FU bolus per 24 hours-period, mEPIC is based on the De Gramont intravenous regimen and consists of administering one intraperitoneal bolus of 5-FU (400 mg/m2) followed by a 24 hours-intraperitoneal infusion of 5-FU (1200 mg/m2) on postoperative days 1 and 2. The total proposed intraperitoneal dose of 1600 mg / m2 per day is comparable to and/or lower than described dosing ranges of 5-FU described in the literature. These doses are equivalent to systemic (intravenous) doses but the systemic exposure would be significantly less due to the known intraperitoneal to plasma area under the curve (AUC) ratios of up to 1000-fold. In this regard, the proposed dose is considered to be toxicologically safe.

The purpose of the study is to confirm the feasibility of mEPIC by evaluating its completion rate compared to the one of historical EPIC cohorts in patients with colorectal and appendicular neoplasms with peritoneal carcinomatosis treated with CRS and HIPEC. The hypothesis of this study is that mEPIC will be superior to the standard EPIC protocol in terms of completion rate. The safety of mEPIC (adverse events) and logistical nursing or pharmaceutical problems will also be recorded and assessed. Demonstrating feasibility of mEPIC will facilitate development of subsequent clinical trials evaluating its efficacy (recurrence free survival) and safety (30-day morbidity/mortality) compared to the standard EPIC protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age 18 years or older, both genders.
* In good general health as evidenced by an ECOG score of 0 or 1.
* Histological diagnosis of appendicular or colorectal tumors with peritoneal carcinomatosis, either synchronous (< 12 months after primary diagnosis) or metachronous (>12 months after the primary diagnosis)
* Complete staging defined as: (1)Computed tomography (CT) scan of the chest, abdomen and pelvis. (2) Positron emission tomography (PET) scan when clinically appropriate. (3) Diagnostic laparoscopy reporting Peritoneal carcinomatosis index (PCI) +/- biopsy
* Meets criteria for recommendation by combined multidisciplinary team and tumor board for cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (CRS+HIPEC) followed by mEPIC
* Surgery must be performed within 4-6 weeks following the end of neoadjuvant therapy or 4-6 weeks following the patient's enrollment if no neoadjuvant therapy needed.
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the study duration
* Hematology: Absolute neutrophil count (ANC) ≥ 1,500/ μL; Platelets > 75,000/ μL.
* Adequate Renal function Creatinine <1.5 x the upper limit of normal (ULN) or calculated creatinine clearance of ≥ 50ml/min.
* Adequate Hepatic function: Bilirubin less than 1.5mg/dL; (except in patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0mg/dL).

Exclusion Criteria:

Pre-cytoreductive surgery:

* Other malignancies other than appendicular and colorectal neoplasms with peritoneal involvement
* Inability to complete cytoreductive surgery (ECOG 2 or above) or any patient deemed unfit for surgery
* Known allergic reaction or major toxicity to Fluorouracil
* Contraindications to Fluorouracil, including history of coronary spasm and/or known dihydropyrimidine dehydrogenase deficiency
* Pregnancy
* Evidence of extensive intraperitoneal adhesions at the time of surgery which prohibits intraperitoneal therapy, as determined by the operating surgeon.
* Any condition that would preclude the ability to deliver appropriate intraperitoneal (IP) therapy.

Post-cytoreductive surgery:

* Patient deemed not medically suitable to receive mEPIC protocol according to surgical team
* Uncorrected coagulopathy and/or thrombocytopenia and/or neutropenia
* Active infection
* Hemodynamic and / or respiratory compromise
* Evidence of extensive intraperitoneal adhesions at the time of surgery which prohibits intraperitoneal therapy, as determined by the operating surgeon.
* Any condition that would preclude the ability to deliver appropriate IP therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of mEPIC | 2 days (assessed at the end of mEPIC protocol).
  Evaluate mEPIC completion rate in patients with colorectal and appendicular cancer with peritoneal carcinomatosis treated with CRS and HIPEC and followed by mEPIC in a tertiary Canadian centre.

SECONDARY OUTCOMES:
Safety of mEPIC | Up to 3 weeks (assessed during the hospitalization following the participant's surgery).
  Evaluate the safety of the mEPIC protocol by monitoring adverse events arising during the protocol.
Satisfaction of care team | 2 days (assessed during mEPIC protocol)
  Assess satisfaction of care team including surgery and nursing teams regarding the implementation process of the mEPIC protocol. It is evaluated using a questionnaire form collecting comments from the care team about logistical barriers encountered during mEPIC protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Soucisse, MD, FRCSC, Principal Investigator — CIUSSS de l'Est-de-l'Île-de-Montréal - Hôpital Maisonneuve-Rosemont
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

REFERENCES:
- [Background] Soucisse ML, Liauw W, Hicks G, Morris DL. Early postoperative intraperitoneal chemotherapy for lower gastrointestinal neoplasms with peritoneal metastasis: a systematic review and critical analysis. Pleura Peritoneum. 2019 Oct 4;4(3):20190007. doi: 10.1515/pp-2019-0007. eCollection 2019 Sep 1. PMID 31667329
- [Background] Cunliffe WJ, Sugarbaker PH. Gastrointestinal malignancy: rationale for adjuvant therapy using early postoperative intraperitoneal chemotherapy. Br J Surg. 1989 Oct;76(10):1082-90. doi: 10.1002/bjs.1800761030. PMID 2688796
- [Background] Sugarbaker PH, Graves T, DeBruijn EA, Cunliffe WJ, Mullins RE, Hull WE, Oliff L, Schlag P. Early postoperative intraperitoneal chemotherapy as an adjuvant therapy to surgery for peritoneal carcinomatosis from gastrointestinal cancer: pharmacological studies. Cancer Res. 1990 Sep 15;50(18):5790-4. PMID 2118420
- [Background] Pestieau SR, Schnake KJ, Stuart OA, Sugarbaker PH. Impact of carrier solutions on pharmacokinetics of intraperitoneal chemotherapy. Cancer Chemother Pharmacol. 2001 Mar;47(3):269-76. doi: 10.1007/s002800000214. PMID 11320672
- [Background] Cashin PH, Mahteme H, Spang N, Syk I, Frodin JE, Torkzad M, Glimelius B, Graf W. Cytoreductive surgery and intraperitoneal chemotherapy versus systemic chemotherapy for colorectal peritoneal metastases: A randomised trial. Eur J Cancer. 2016 Jan;53:155-62. doi: 10.1016/j.ejca.2015.09.017. Epub 2016 Jan 2. PMID 26751236
- [Background] Huang Y, Alzahrani NA, Liauw W, Traiki TB, Morris DL. Early Postoperative Intraperitoneal Chemotherapy for Low-Grade Appendiceal Mucinous Neoplasms with Pseudomyxoma Peritonei: Is it Beneficial? Ann Surg Oncol. 2017 Jan;24(1):176-183. doi: 10.1245/s10434-016-5529-0. Epub 2016 Oct 7. PMID 27718032
- [Background] Lam JY, McConnell YJ, Rivard JD, Temple WJ, Mack LA. Hyperthermic intraperitoneal chemotherapy + early postoperative intraperitoneal chemotherapy versus hyperthermic intraperitoneal chemotherapy alone: assessment of survival outcomes for colorectal and high-grade appendiceal peritoneal carcinomatosis. Am J Surg. 2015 Sep;210(3):424-30. doi: 10.1016/j.amjsurg.2015.03.008. Epub 2015 May 12. PMID 26051744
- [Background] Hayler R, Lockhart K, Barat S, Cheng E, Mui J, Shamavonian R, Ahmadi N, Alzahrani N, Liauw W, Morris D. Survival benefits with EPIC in addition to HIPEC for low grade appendiceal neoplasms with pseudomyxoma peritonei: a propensity score matched study. Pleura Peritoneum. 2023 Mar 16;8(1):27-35. doi: 10.1515/pp-2022-0205. eCollection 2023 Mar. PMID 37020474
- [Background] Van der Speeten K, Govaerts K, Stuart OA, Sugarbaker PH. Pharmacokinetics of the perioperative use of cancer chemotherapy in peritoneal surface malignancy patients. Gastroenterol Res Pract. 2012;2012:378064. doi: 10.1155/2012/378064. Epub 2012 Jun 13. PMID 22778722
- [Background] Jacquet P, Averbach A, Stephens AD, Stuart OA, Chang D, Sugarbaker PH. Heated intraoperative intraperitoneal mitomycin C and early postoperative intraperitoneal 5-fluorouracil: pharmacokinetic studies. Oncology. 1998 Mar-Apr;55(2):130-8. doi: 10.1159/000011847. PMID 9499187
- [Background] Meta-analysis Group In Cancer; Piedbois P, Rougier P, Buyse M, Pignon J, Ryan L, Hansen R, Zee B, Weinerman B, Pater J, Leichman C, Macdonald J, Benedetti J, Lokich J, Fryer J, Brufman G, Isacson R, Laplanche A, Levy E. Efficacy of intravenous continuous infusion of fluorouracil compared with bolus administration in advanced colorectal cancer. J Clin Oncol. 1998 Jan;16(1):301-8. doi: 10.1200/JCO.1998.16.1.301. PMID 9440757
- [Background] Thomas DM, Zalcberg JR. 5-fluorouracil: a pharmacological paradigm in the use of cytotoxics. Clin Exp Pharmacol Physiol. 1998 Nov;25(11):887-95. doi: 10.1111/j.1440-1681.1998.tb02339.x. PMID 9807659
- [Background] Muggia FM, Chan KK, Russell C, Colombo N, Speyer JL, Sehgal K, Jeffers S, Sorich J, Leichman L, Beller U, et al. Phase I and pharmacologic evaluation of intraperitoneal 5-fluoro-2'-deoxyuridine. Cancer Chemother Pharmacol. 1991;28(4):241-50. doi: 10.1007/BF00685529. PMID 1831736
- [Background] Oman M, Lundqvist S, Gustavsson B, Hafstrom LO, Naredi P. Phase I/II trial of intraperitoneal 5-Fluorouracil with and without intravenous vasopressin in non-resectable pancreas cancer. Cancer Chemother Pharmacol. 2005 Dec;56(6):603-9. doi: 10.1007/s00280-005-1012-5. Epub 2005 Jul 27. PMID 16047145
- [Background] Kerr DJ, Young AM, Neoptolemos JP, Sherman M, Van-Geene P, Stanley A, Ferry D, Dobbie JW, Vincke B, Gilbert J, el Eini D, Dombros N, Fountzilas G. Prolonged intraperitoneal infusion of 5-fluorouracil using a novel carrier solution. Br J Cancer. 1996 Dec;74(12):2032-5. doi: 10.1038/bjc.1996.672. PMID 8980409